CLINICAL TRIAL: NCT03051009
Title: A Multi-Centre Trial Investigating the Long Term Safety and Tolerability of Desmopressin (FE 992026) Orally Disintegrating Tablets for the Treatment of Nocturia Due to Nocturnal Polyuria in Japanese Subjects
Brief Title: Trial Investigating the Long Term Safety and Tolerability of Desmopressin Orally Disintegrating Tablets (ODT) for Nocturia Due to Nocturnal Polyuria in Japanese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000131
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Intervention Model Description: The trial is designed as partly an extension trial for subjects completing trial 000129 (female subjects) and 000130 (male subjects) and partly as a trial for new female and male subjects.
Who Masked: Participant, Investigator
Masking Description: One dose level (25 μg desmopressin OCD) is included for female subjects and will be open-labelled for all female subjects.
  Two different dose levels (25 μg desmopressin and 50 μg desmopressin ODT are included for male subjects in a double-blinded manner. Male subjects continuing from trial 000130 will continue their randomised treatment and subjects who received placebo will be randomised to one of the 2 dose levels (25 μg desmopressin or 50 μg desmopressin ODT).
  New male subjects will be allocated to receive 50 μg desmopressin ODT in an open-labelled manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Desmopressin ODT 25 μg (female previous on 25 μg) (Experimental): Subjects received 25 μg in trial 000129.
  Interventions: Drug: Desmopressin ODT 25 μg
- Desmopressin ODT 25 μg (female previously on placebo) (Experimental): Subjects received placebo in trial 000129
  Interventions: Drug: Desmopressin ODT 25 μg
- Desmopressin ODT 25 μg (female) (Experimental): New female subjects
  Interventions: Drug: Desmopressin ODT 25 μg
- Desmopressin ODT 25 μg (male previous on 25 μg) (Experimental): Subjects received 25 μg in trial 000130
  Interventions: Drug: Desmopressin ODT 25 μg
- Desmopressin ODT 50 μg (male previous on 50 μg) (Experimental): Subjects received 50 μg in trial 000130
  Interventions: Drug: Desmopressin ODT 50 μg
- Desmopressin ODT 50 μg (male previous on placebo) (Experimental): Subjects received placebo in trial 000130
  Interventions: Drug: Desmopressin ODT 50 μg
- Desmopressin ODT 25 μg (male) (Experimental): Subjects received placebo in trial 000130
  Interventions: Drug: Desmopressin ODT 25 μg
- Desmopressin ODT 50 μg (male) (Experimental): New male subjects
  Interventions: Drug: Desmopressin ODT 50 μg

INTERVENTIONS:
Drug: Desmopressin ODT 25 μg
  Other Names: FE 992026
  Arms: Desmopressin ODT 25 μg (female previous on 25 μg); Desmopressin ODT 25 μg (female previously on placebo); Desmopressin ODT 25 μg (female); Desmopressin ODT 25 μg (male previous on 25 μg); Desmopressin ODT 25 μg (male)
Drug: Desmopressin ODT 50 μg
  Other Names: FE 992026
  Arms: Desmopressin ODT 50 μg (male previous on 50 μg); Desmopressin ODT 50 μg (male previous on placebo); Desmopressin ODT 50 μg (male)

SUMMARY:
Demonstrate the safety and tolerability of desmopressin ODT during long-term treatment of subjects with nocturia due to nocturnal polyuria, for up to 1 year

ELIGIBILITY:
Inclusion Criteria (for subjects who participated in trials 000129 or 000130):

* Written informed consent prior to performance of any trial-related activity for the 000131 trial
* Has completed participation in trial 000129 or 000130

Exclusion Criteria (for subjects who participated in trials 000129 or 000130):

* Hyponatraemia (serum sodium level <135 mmol/L) at Visit 7 in trial 000129 or 000130
* Withdrawal from clinical trial 000129 or 000130

Inclusion Criteria (for subjects who did not participate in trials 000129 or 000130):

* Written informed consent prior to performance of any trial-related activity
* Adult ≥20 years of age
* Nocturia symptoms present for ≥6 months prior to trial entry at Visit 1a
* Nocturnal polyuria at the end of screening period prior to Visit 1b
* Bothered by nocturia on the Hsu 5-point Likert bother scale at Visit 1a and Visit 1b
* Has given agreement about contraception during the trial

Exclusion Criteria (for subjects who did not participate in trials 000129 or 000130):

* Early withdrawal from clinical trial 000129 or 000130
* Evidence of any significant voiding dysfunction resulting in abnormally low bladder capacity at the end of the screening period prior to Visit 1b
* History or evidence of significant obstructive sleep apnoea
* History or diagnosis of any of the following urological diseases:

  * Interstitial cystitis or bladder pain disorder
  * In males, suspicion of moderate or severe benign prostate hyperplasia (BPH), defined as international prostate symptom score (IPSS) ≥8 points and:

    * Urinary flow <5 mL/s or
    * Post-void residual volume >150 mL
  * Stress urinary incontinence or mixed incontinence, where stress incontinence is the predominant component based on prior history
  * Chronic prostatitis/chronic pelvic pain syndrome
* Surgical treatment, including transurethral resection, for BOO or BPH within the past 6 months prior to Visit 1a
* Symptoms of severe over-active bladder (OAB):

  * Defined as an over-active bladder symptom score (OABSS) ≥12 at Visit 1a
  * Defined as a mean of >8 voids and a mean of ≥1 urgency episode per 24 hours at the end of the screening period prior to Visit 1b
* Genito-urinary tract pathology that can in the investigator's opinion be responsible for urgency or urinary incontinence at Visit 1a
* Complication of cancer or a history of cancer which has not been in remission for the last 5 years at Visit 1a
* Current or a history of urologic malignancies, any lower urinary tract surgery, previous pelvic irradiation, or neoplasia at Visit 1a
* History of any neurological disease affecting bladder function or muscle strength at Visit 1a
* Habitual or psychogenic polydipsia based on medical history at Visit 1a or 24-hour urine output of >2.8 L based on the voiding diary at Visit 1b
* Central or nephrogenic diabetes insipidus at Visit 1a
* Syndrome of inappropriate antidiuretic hormone secretion at Visit 1a
* Suspicion or evidence of cardiac failure at Visit 1a
* Uncontrolled hypertension at Visit 1a and Visit 1b
* Hyponatraemia (serum sodium level <135 mmol/L) at Visit 1a Renal insufficiency at Visit 1a and Visit 1b
* Renal insufficiency at Visit 1a and Visit 1b
* Hepatic and/or biliary diseases at Visit 1a and Visit 1b
* Known or suspected hypersensitivity to desmopressin ODTs or previous desmopressin treatment for nocturia at Visit 1a
* In females, pregnancy, breastfeeding, or a plan to become pregnant during the period of the clinical trial.
* Known alcohol or substance abuse at Visit 1a
* Work or lifestyle that may interfere with regular night-time sleep at Visit 1a, e.g., shift workers
* Any other medical condition, laboratory abnormality, psychiatric condition, mental incapacity, or language barrier that, in the judgment of the investigator, would impair participation in the trial at Visit 1a
* Use of any prohibited therapy during the trial period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of adverse events | Up to 1 year
  During long-term treatment
Clinically significant changes in laboratory values and vital signs | Up to 1 year
  During long-term treatment
The incidence and severity of hyponatraemia | Up to 1 year
  Measured by serum sodium levels during long-term treatment

SECONDARY OUTCOMES:
Change from baseline in mean number of nocturnal voids | Week 12, 24, 40 and 52
Change from baseline in mean time to first awakening to void | Week 12, 24, 40 and 52
Change from baseline in mean nocturnal urin volume | Week 12, 24, 40 and 52
Change from baseline in mean Nocturnal Polyuria Index (NPI) | Week 12, 24, 40 and 52
Change from baseline in Nocturia-Specific Quality-of-Life Questionnaire (N-QoL) | Week 12, 24, 40 and 52
Change from baseline in Insomnia Severity Index (ISI) | Week 12, 24, 40 and 52
Change from baseline in bother score | Week 12, 24, 40 and 52
  Assessed by the Hsu 5-point Likert bother scale

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Investigational site (there may be other sites in this country), Tokyo, Japan